CLINICAL TRIAL: NCT02373241
Title: Chronobiology and Chronopharmacology to Prevent Sickle Cell Kidney Disease
Brief Title: Preventing Sickle Cell Kidney Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Estimated GFR was determined not to be a reliable endpoint for this study. We identified significant variabilty in annual eGFR that it became inappropriate to randomize to a medication but use EGFR as the primary endpoint.
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey D. Lebensburger, DO, Assistant Professor of Pediatric Hematology Oncology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F141107009; 1K23HL127100-01 (NIH)
Record Dates: First submitted 2015-02-05; First posted 2015-02-26 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Anemia, Sickle Cell; Sickle Cell Disease; Kidney Disease; Hypertension; Proteinuria
Keywords: Anemia, Sickle Cell; Sickle Cell Disease; Kidney Disease; Hypertension; Proteinuria; Losartan; Antihypertensive Agents; Blood Pressure
MeSH Terms: conditions — Anemia, Sickle Cell; Kidney Diseases; Hypertension; Proteinuria | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Blood Pressure Management (Active Comparator): Participants initiated on 25mg of losartan daily and randomized to lower in-clinic BP to <95th percentile
  Interventions: Drug: Losartan
- Experimental Blood Pressure Management (Experimental): Participants initiated on 25mg of losartan daily and randomized to lower in-clinic BP to <75th percentile
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — Standard dosing
  Other Names: coozar
  Arms: Standard Blood Pressure Management
Drug: Losartan — Experimental dosing
  Other Names: coozar
  Arms: Experimental Blood Pressure Management

SUMMARY:
Untreated hypertension and renal injury are risk factors for increased morbidity and mortality in sickle cell disease, yet early markers of progressive disease have not been identified and therapies to prevent the development of adverse cardiovascular outcomes have not been defined. Circadian blood pressure, as defined by 24 hour blood pressure monitoring, is more accurate than clinic blood pressure in defining secondary hypertension and abnormal nocturnal blood pressured dipping and nocturnal hypertension have been linked to progressive renal disease in other diseases.

Methodology/Aims: A randomized feasibility trial of losartan will be conducted among adolescent HbSS and SB0 thalassemia patients (11-19 years) with abnormal nocturnal blood pressure dipping. During this six month feasibility trial, two dosing strategies of losartan (titrated to keep clinic BP <95th percentile vs. <75th percentile) will be analyzed for safety and effect on restoring normal circadian blood pressure.

A prospective cohort study among HbSS and SB0 thalassemia patients (6-19 years) will also be conducted to evaluate the incidence of hypertension and role of monitoring potential biomarkers of kidney injury and hypertension. Cohort participants will undergo annual evaluations of hypertension(24 hour blood pressure monitoring for participants ≥ 11yrs, clinic BP in all participants) and markers of kidney injury/hypertension.

Expected Results: At the completion of the feasibility trial, vital background information will be obtained to design a definitive multicenter trial of hypertension in sickle cell disease. At the completion of the cohort study, the incidence of pediatric hypertension will be identified and the role for monitoring blood and urine biomarkers will be better understood.

As therapy for patients with renal failure is dismal, it is imperative that SCD patients at risk are identified early and that therapeutic trials are conducted that prevent progression.

DETAILED DESCRIPTION:
Feasibility Trial of Losartan to Correct Abnormal Circadian Blood Pressure. Cohort participants (below) identified with in-clinic hypertension and abnormal nocturnal dipping on 24 hour ABPM will be asked to participate in a feasibility trial of losartan. Participants will be offered a consultation with Pediatric Nephrology prior to study enrollment. Participants that consent /assent will undergo repeat 24 hour ABPM to confirm abnormal circadian blood pressure prior to receiving losartan. At baseline, participants will undergo evaluation for biomarkers of kidney injury and hypertension. Participants will start on losartan at 25mg of losartan and randomized to titrate clinic BP <95th or 75th percentile based on NHLBI BP tables. Participants will be followed monthly x 6 months and receive standard of care labs. ABPM and blood/urine biomarkers of kidney injury, buccal swab for circadian genes, and hypertension will be repeated at 3 and 6 months. Participants will undergo monthly evaluation for adherence through pill counting and questionnaires. Safety of dosing will be monitored by internal review and external review (DSMB).

Prospective Pediatric Cohort to Evaluate Hypertension and Kidney Injury. Patients with HbSS or SB0 thalassemia, ages ≥ 6 years and have signed informed consent will undergo clinic BP, annual ABPM and biomarkers to determine the incidence of HTN and potential role for biomarkers as monitors for the development of hypertension or kidney injury/disease. Urine will be collected annually and evaluated for current known biomarkers of kidney disease and stored for future analysis of relevant biomarkers. Uric acid will be processed from collected blood annually.

ELIGIBILITY:
Inclusion Criteria:

* Pts with HbSS or SB0 thalassemia
* Hypertension from clinic BP readings (defined by NHLBI BP tables)
* Abnormal nocturnal dipping (systolic or diastolic) as defined by <10% dip or abnormal nocturnal BP load (>25% of sleep BP readings >95th percentile as defined by AHA ABPM guidelines)
* Signed Informed Consent

Exclusion Criteria:

* Patient already on BP lowering medication
* Hyperkalemia
* Pregnancy

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2015-04; Primary Completion 2021-02 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Lebensburger, DO, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Samuels J, Ng D, Flynn JT, Mitsnefes M, Poffenbarger T, Warady BA, Furth S; Chronic Kidney Disease in Children Study Group. Ambulatory blood pressure patterns in children with chronic kidney disease. Hypertension. 2012 Jul;60(1):43-50. doi: 10.1161/HYPERTENSIONAHA.111.189266. Epub 2012 May 14. PMID 22585950
- [Background] Seeman T, Palyzova D, Dusek J, Janda J. Reduced nocturnal blood pressure dip and sustained nighttime hypertension are specific markers of secondary hypertension. J Pediatr. 2005 Sep;147(3):366-71. doi: 10.1016/j.jpeds.2005.04.042. PMID 16182677
- [Background] Okuguchi T, Osanai T, Fujiwara N, Kato T, Metoki N, Konta Y, Okumura K. Effect of losartan on nocturnal blood pressure in patients with stroke: comparison with angiotensin converting enzyme inhibitor. Am J Hypertens. 2002 Nov;15(11):998-1002. doi: 10.1016/s0895-7061(02)02998-9. PMID 12441222
- [Background] Flynn JT, Daniels SR, Hayman LL, Maahs DM, McCrindle BW, Mitsnefes M, Zachariah JP, Urbina EM; American Heart Association Atherosclerosis, Hypertension and Obesity in Youth Committee of the Council on Cardiovascular Disease in the Young. Update: ambulatory blood pressure monitoring in children and adolescents: a scientific statement from the American Heart Association. Hypertension. 2014 May;63(5):1116-35. doi: 10.1161/HYP.0000000000000007. Epub 2014 Mar 3. No abstract available. PMID 24591341
- [Background] Lebensburger JD, Palabindela P, Howard TH, Feig DI, Aban I, Askenazi DJ. Prevalence of acute kidney injury during pediatric admissions for acute chest syndrome. Pediatr Nephrol. 2016 Aug;31(8):1363-8. doi: 10.1007/s00467-016-3370-0. Epub 2016 Mar 24. PMID 27011218
- [Background] Aban I, Baddam S, Hilliard LM, Howard TH, Feig DI, Lebensburger JD. Severe anemia early in life as a risk factor for sickle-cell kidney disease. Blood. 2017 Jan 19;129(3):385-387. doi: 10.1182/blood-2016-09-738104. Epub 2016 Dec 5. No abstract available. PMID 27919909
- [Background] Baddam S, Aban I, Hilliard L, Howard T, Askenazi D, Lebensburger JD. Acute kidney injury during a pediatric sickle cell vaso-occlusive pain crisis. Pediatr Nephrol. 2017 Aug;32(8):1451-1456. doi: 10.1007/s00467-017-3623-6. Epub 2017 Feb 25. PMID 28238158
- [Background] Lebensburger JD, Cutter GR, Howard TH, Muntner P, Feig DI. Evaluating risk factors for chronic kidney disease in pediatric patients with sickle cell anemia. Pediatr Nephrol. 2017 Sep;32(9):1565-1573. doi: 10.1007/s00467-017-3658-8. Epub 2017 Apr 5. PMID 28382567
- [Background] Lebensburger JD, Aban I, Hilliard LM, Feig DI. Hyperuricemia and abnormal nocturnal dipping impact glomerular filtration rate in patients with sickle cell anemia. Am J Hematol. 2021 May 1;96(5):E143-E146. doi: 10.1002/ajh.26115. Epub 2021 Feb 18. No abstract available. PMID 33524174

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Blood Pressure Management | Experimental Blood Pressure Management
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 patient identified as eligible for the study due to ambulatory hypertension
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Blood Pressure Management | Experimental Blood Pressure Management | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 1 | 1
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] |  | 16 [16 to 16] | 16 [16 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 1 | 1
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by the Number of Patients That Accept Enrollment, Remain Adherent to Losartan, and Remain Adherent to Study Procedures.
Description: Outcome 1a. Document the rate of acceptance (quantitative) and reasons for acceptance/rejection (qualitative) in a randomized trial of trial of losartan for SCD patients with abnormal nocturnal blood pressures.
  Outcome 1b. Identify the adherence rate to losartan during a randomized three year trial of losartan for SCD patients (n=40) with abnormal nocturnal blood pressure.
  Outcome 1c. Determine the adherence rate to study procedures among participants enrolled in a three year trial of losartan for SCD patients (n=40) with abnormal nocturnal blood pressure.
Time Frame: 5 yrs
Population: We stopped the RCT as eGFR was determined not to be an accurate measure of GFR in SCD patients
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Blood Pressure Management | Experimental Blood Pressure Management
Number analyzed (Participants) | 0 | 1
Participants | 0 | 1

2. Secondary Outcome: Number of Patients With Incident Hypertension
Description: We will prospectively evaluate the incidence of hypertension (Clinic BP in pts >5yrs and ABPM in pts >10 yrs) and role of blood and urine biomarkers (pts >5ys) among participants with HbSS or SB0 thalassemia (expected cohort n=200) over 5 yrs. We identified 20 participants (34%) with incident hypertension but randomized one to the study. The study was terminated as the eGFR was determined not to be a reliable endpoint in pediatric sickle cell.
Time Frame: 5 yrs
Population: This study was terminated early so we did not perform analysis of losartan on incident hypertension.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Blood Pressure Management | Experimental Blood Pressure Management
Number analyzed (Participants) | 0 | 1
Participants | 0 | 1

3. Secondary Outcome: Feasibility as Measured by the Number of Patients With Improvement in Nocturnal Blood Pressure While Receiving Losartan.
Description: As a feasibility trial, the effect of losartan on lowering nocturnal hypertension will be monitored to identify the difference in nocturnal BP improvement between the two treatment arms, and within group standard deviation of BP
Time Frame: 5 years
Population: We did not have any patients randomized to standard blood pressure management
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Blood Pressure Management | Experimental Blood Pressure Management
Number analyzed (Participants) | 0 | 1
Participants |  | 1

ADVERSE EVENTS:
Time Frame: 5 years
Description: No adverse events reported
Arm/Group | Standard Blood Pressure Management | Experimental Blood Pressure Management
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT02373241/Prot_SAP_000.pdf